CLINICAL TRIAL: NCT00783809
Title: Measurement of Optic Nerve Sheath in Traumatic Raised Intracranial Pressure
Acronym: MOONSTRIP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Niv Sne, Director of Trauma Research, McMaster University
Other Study IDs: PSI-34-2008
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Traumatic Brain Injury
Keywords: intracranial pressure; intracranial hypertension; ultrasound; emergency; traumatic brain injury; ocular ultrasound
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Trauma patients are at risk for serious head trauma. The consequences of serious head trauma are often life altering. Currently, the only method available to rapidly assess the severity of head injury and need for neurosurgical intervention is the CT scan. This time consuming test requires transportation of a potentially unstable patient to the CT scanner.

The investigators goal in traumatic brain injury is to identify early those patients who may require neurosurgical intervention. Brain swelling (elevated intracranial pressure) is transmitted to the eye and this can be measured with ultrasound. The investigators hypothesis is that this test will rule out significant elevations in intracranial pressure and perform as well as CT scan in doing this.

The investigators study aims to demonstrate that ultrasound of the optic nerve is as good as CT scan in ruling out clinically significant elevations in pressure within the brain. After consent has been obtained, any trauma patient who has an indication to undergo CT scan of the brain will also undergo ultrasound of the eye. A radiologist will then review the CT scans to determine if signs of elevated intracranial pressure are present. The investigators hope to demonstrate that a bedside ultrasound performed in the trauma suite is reliable for ruling out the possibility of elevated intracranial pressure.

**Update August 2009** Currently, deferred consent has been obtained from our REB allowing us to defer consent for this intervention of minimal risk. As well, REB has also approved phone consent in the interim.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 16 involved in blunt trauma.
* Patient is to undergo a CT of the head to evaluate suspected closed head injury
* Consent and ultrasound can be preformed within 1 hour before or after CT of the head

Exclusion Criteria:

* Penetrating trauma to the head or significant ocular trauma
* Patients not expected to survive transfer out of the emergency room department
* Patient is too unstable to undergo a CT of the head or ultrasound of the optic nerve

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who present to the emergency department with suspected closed head injury as a result of blunt trauma and require CT head
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Elevation in intracranial pressure as estimated by CT scan or ICP monitor | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Niv Sne, MD FRCSC, Principal Investigator — Hamilton Health Sciences Corporation; Andrew J Healey, MD FRCPC, Study Chair — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Koziarz A, Sne N, Kegel F, Alhazzani W, Nath S, Badhiwala JH, Rice T, Engels P, Samir F, Healey A, Kahnamoui K, Banfield L, Sharma S, Reddy K, Hawryluk GWJ, Kirkpatrick AW, Almenawer SA. Optic nerve sheath diameter sonography for the diagnosis of increased intracranial pressure: a systematic review and meta-analysis protocol. BMJ Open. 2017 Aug 11;7(8):e016194. doi: 10.1136/bmjopen-2017-016194. PMID 28801417